CLINICAL TRIAL: NCT06323681
Title: A Prospective, Multicenter, Non-randomized, Controlled Study to Pursuit Clinical Functional Cure of Pegylated Interferon α in Previously Interferon-treated Chronic Hepatitis B （Leading Study）
Brief Title: Pegylated Interferon α in Previously Interferon-treated CHB（Leading Study）
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qing XIe (Other)
Responsible Party: Sponsor-Investigator, Qing XIe, Director of Department of Infectious Disease, Rui Jin, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Leading Study
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Hepatitis b
Keywords: CHB, peginterferon, functional cure, retreatment
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peginterferon α-2b based treatment group (Experimental)
  Interventions: Drug: Peginterferon α-2b based treatment group
- NAs monotherapy group (Active Comparator)
  Interventions: Drug: NAs monotherapy group

INTERVENTIONS:
Drug: Peginterferon α-2b based treatment group — Peginterferon α-2b injection, 180mcg, s.c, once a week, for 48 weeks. If the baseline HBV DNA is higher than the minimum detection limit (using high-sensitivity kit), combined with nucleos(t)ide analogs (NAs) is recommended.
  Arms: Peginterferon α-2b based treatment group
Drug: NAs monotherapy group — First-line NAs (e.g. Entecavir (ETV), tenofovir disoproxil fumarate (TDF), tenofovir alafenamide fumarate (TAF), tenofovir amibufenamide (TMF)), one tablet a day, take orally, for 48 weeks.
  Arms: NAs monotherapy group

SUMMARY:
Previous clinical practice and exploratory studies suggest that some patients who have not achieved functional cure in the first round of interferon therapy can achieve HBsAg clearance by interferon retreatment (intermittent therapy), which can reduce the occurrence of complications such as liver fibrosis, liver cirrhosis and liver cancer, and its clinical benefit is expected to be higher than that of NAs monotherapy.

This study is aimed to conduct a large-scale, multicenter, prospective study to confirm the benefit of peginterferon-based therapies in these populations. It expected to enroll about 2000 patients with chronic hepatitis B who have received prior interferon therapy and achieved a good response but without function cure, patients receive either interferon-based therapy or NAs monotherapy, according to their wishes and doctors' professional recommendations, with a ratio of 2:1 between the two groups, and all patients treated for 48 weeks. The HBsAg clearance rate before and after treatment, safety, etc. will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign the informed consent, participate in the study voluntarily.
* Aged between 18 and 65 (including 18 and 65).
* HBsAg positive for at least 6 months or other evidence suggests chronic hepatitis B.
* Had previously received interferon therapy, and discontinuation for at least 6 months at the time of enrollment, with a HBsAg level declined for at least 80% at the end of interferon treatment compared to the level of treatment started.
* HBsAg≤500 IU/mL at screening, and HBsAg rebound should not exceed 50% when compared to the HBsAg level of previously interferon treatment started.
* The pregnancy test within 24 hours previous to the first medication must be negative for women of childbearing. And all participants (male and female) should use effective contraception during the study period.

Exclusion Criteria:

* Pregnant or lactating women, or those who had a birth plan during the study period.
* Patients with neuropsychiatric disorders, especially depression, anxiety, mania, schizophrenia and other mental illness history or family history of mental illness.
* Patients with chronic liver disease caused by hepatitis A, hepatitis C, hepatitis E and/or HIV infection, or other causes (such as alcoholic hepatitis, drug-induced hepatitis, autoimmune liver disease, etc.).
* Evidence of acute severe liver damage: ALT>10 ULN, or markedly elevated ALT with significantly elevated bilirubin.
* Evidence of uncompensated liver disease: ascites, esophageal and gastric varices rupture bleeding, sepsis, hepatic encephalopathy, hepatorenal syndrome, etc. Or previous evidence of decompensation of cirrhosis.
* Patients with evidence of hepatocellular carcinoma or AFP>1 ULN.
* Kidney diseases: acute or chronic nephritis, renal insufficiency, nephrotic syndrome, etc. Or serum creatinine >1 ULN at screening.
* Neutrophil count <1.5×10^9/L, platelet count <90×10^9/L, blood phosphorus < 0.8 mmol /L.
* Autoimmune diseases (such as psoriasis, systemic erythematosus, etc.), endocrine system diseases (such as thyroid diseases, diabetes, etc.), hypertension (blood pressure ≥140/90 mmHg) poorly controlled by prescription drugs, serious history of heart disease (especially in the past 6 months), severe retinopathy or other serious eye diseases. Patients with organic disease or dysfunction of other vital organs.
* Patients who plan to receive organ transplant or have already undergone organ transplant.
* Patients who allergic to the investigational drug or any of its excipients, or who meet any contraindication declared in the instructions of the investigational drug.
* Other conditions that are considered inappropriate for enrollment by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2016 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with HBsAg below the lower limit of detection. | Week 48

SECONDARY OUTCOMES:
Decrease of HBV DNA levels at week 48 compared to baseline. | Week 48
Proportion of patients with HBV DNA below the lower limit of detection. | Week 48
Decrease of HBsAg levels at week 48 compared to baseline. | Week 48
Proportion of patients with HBsAg seroconversion. | Week 48
Proportion of patients with HBeAg below the lower limit of detection for patients with baseline HBeAg positive. | Week 48
Proportion of patients with HBeAg seroconversion for patients with baseline HBeAg positive. | Week 48
Serious adverse events. | from baseline to 48 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases , Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China